Official title: Physical Therapy Intervention for Puerperal Mastitis

Number: NCT04569136

Document date: 04/01/2022

Introduction

Puerperal mastitis is one of the most commonly reported problems during

breastfeeding (1-3). Women frequently report breast pain, tenderness, redness,

engorgement, fever, malaise, chills, lethargy, sweating, headache, nipple damage and

a hot spot on the affected breast (4-6). These highly distressing symptoms may

severely impact on a woman's daily activities and quality of life and might lead to the

premature cessation of exclusive breastfeeding, which may have significant impact on

infant health and survival.

The role of physical therapy in reducing pregnancy/postpartum-related disorders

including breast problems is gaining momentum and importance in obstetrics (7).

However, to date, only low-level evidence has shown positive effects of breast

massage, a physical technique, on pain, milk supply and symptom relief in women

with breastfeeding problems (7). This is encouraging, however further research is

needed to explore whether physical therapy is effective to reduce symptoms of

1

puerperal mastitis. Therefore, the aims of this study were to explore clinical effects of therapeutic ultrasound, education and massage on mastitis symptoms and to compare the effectiveness of therapeutic ultrasound, education and massage versus usual obstetric care and sham ultrasound treatment on patient-centered outcomes in the short- and medium-term.

## Methods

A randomized controlled trial was conducted from May 2021 to April 2023.

Postpartum lactating women aged from 21 to 45 with breast symptoms were recruited through the Obstetrics and Gynecology Clinic of National Cheng Kung University

Hospital, the postpartum care centers, websites and community. Eligible participants were randomly allocated to the ultrasound group, sham group, or usual care group.

Participants allocated to the 'Ultrasound' arm of the trial participated in four one-hour treatment sessions with the physical therapist over one week. The treatment included educating the patient about mastitis and self-management strategies, treating with therapeutic ultrasound and administering and teaching breast massage. Participants allocated to the 'Sham' group received the same education and breast massage sessions as described above. In addition, the sham control group received 5 minutes of 'sham' ultrasound at 0 W/cm2 intensity from a physical therapist. Participants

allocated to the 'Usual care' group received usual obstetric care, which included verbal advice/printed patient information regarding mastitis and breastfeeding from the medical or nursing staff. The outcome measures including severity of breast symptoms (breast and nipple pain, breast engorgement), breast hardness, body temperature, breast temperature, breastfeeding self-efficacy, and milk volume were assessed at baseline, immediately post-intervention, and at 3 months following baseline. The acceptability of the intervention program and adverse events were recorded immediately post-intervention and at 3 months following baseline.

## Statistical analysis plan

The data were analyzed using intention-to-treat principles with the SPSS version 20.0 for Windows. The last observation carried forward imputation was used for imputing missing data. Descriptive statistics were used to summarize and report data. All outcome data were assessed for normality using the Kolmogorov-Smirnov test.

Repeated measures analysis of variance with Bonferroni post hoc comparisons was used to compare changes in outcome variables between groups. The equivalent non-parametric tests (i.e. Friedman test and Kruskal Wallis test) were used if data were not normally distributed. Numbers, percentages, mean, standard deviation, median, interquartile range, and p-values were reported. All analyses were tested with a

significance level of p<0.05.

## References

- Scott JA, Robertson M, Fitzpatrick J, Knight C, Mulholland S. Occurrence of lactational mastitis and medical management: a prospective cohort study in Glasgow. Int Breastfeed J. 2008;3:21.
- Amir LH, Forster DA, Lumley J, McLachlan H. A descriptive study of mastitis
  in Australian breastfeeding women: incidence and determinants. BMC Public
  Health. 2007;7:62.
- 3. Kinlay JR, O'Connell DL, Kinlay S. Incidence of mastitis in breastfeeding women during the six months after delivery: a prospective cohort study. Med J Aust. 1998;169(6):310-2.
- Cusack L, Brennan M. Lactational mastitis and breast abscess diagnosis and management in general practice. Aust Fam Physician. 2011;40(12):976-9.
- 5. Ezrati JB, Gordon H. Puerperal mastitis: causes, prevention, and management. J
  Nurse Midwifery. 1979;24(6):3-8.
- 6. Foxman B, D'Arcy H, Gillespie B, Bobo JK, Schwartz K. Lactation mastitis: occurrence and medical management among 946 breastfeeding women in the United States. Am J Epidemiol. 2002;155(2):103-14

7. Mangesi L, Zakarija-Grkovic I. Treatments for breast engorgement during lactation. Cochrane Database Syst Rev. 2016(6):CD006946.